CLINICAL TRIAL: NCT02154945
Title: Retinal Nerve Fiber Layer and Macular Thickness Changes During Pregnancy by Optical Coherence Tomography: Prospective, Observational, Nonrandomized Controlled Study
Brief Title: Retinal Nerve Fiber Layer and Macular Thickness Changes During Pregnancy
Status: Withdrawn | Type: Observational
Why Stopped: Did not go through with the study for logistical reasons
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Other Study IDs: 33-2013.CTIL
Record Dates: First submitted 2014-05-28; First posted 2014-06-04 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2014-06

CONDITIONS: Pregnancy; Retinal Nerve Fiber Layer Thickness; Macular Thickness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose:

Primary: to prospectively measure Retinal Nerve Fiber Layer (RNFL) and macular thickness changes during pregnancy by Optical coherence tomography

Secondary: The effect of pregnancy abnormalities on RNFL and macular thickness in participants who develop systemic or ocular complications during the study period.

DETAILED DESCRIPTION:
There are several known ophthalmic physiologic changes in pregnancy:

1. Refractive Change: progesterone-mediated changes in fluid content partially accounts for refractive change of lens and cornea; myopic shift of less than 1 D was observed in in 15% of participating pregnant women
2. Night vision decreased mainly with low serum vitamin A levels in pregnant women.
3. Fall of the IOP in second half of pregnancy (about 10% drop)
4. Corneal changes (increased thickness; decreased sensitivity) = contact lens intolerance

The retina and optic nerve are considered part of central nervous system, the retina and choroid are highly vascularized. Due to changes in CSF and brain volume, vascular and fluid changes all over the pregnant woman's body we expect to find changes in RNFL and macular thickness during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 1st trimester (6-14w) pregnant healthy women
* No known medical problems related to their current pregnancy on recruitment
* Age 18-45yrs
* No known retinal or optic nerve disease
* Refraction between +3.0 and -4.0 diopters
* Agrees to participate in the study

Exclusion Criteria:

* Retinal or optic nerve disease
* Refractive errors more than +3.0 and -4.0.
* If already finished 14w gestation when recruited to the 1st OCT examination
* Known to have HTN or DM before gestation
* Ocular media abnormality that obscures OCT view or examination

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Retinal nerve fiber layer(RNFL) and Macular thickness by Optical coherence tomography(OCT) during pregnancy | 1 year
  The RNFL, measured in micrometers, will be followed up during the study. Every trimester (starting at the 1st trimester) an OCT will be performed measuring the thickness of the RNFL.
  An OCT will be performed 3 months postpartum as a control.
  The Macular thickness will be measured in the same manner.

SECONDARY OUTCOMES:
Effect of systemic and ocular diseases on Retinal Fiber Layer and Macula during pregnancy | 1 year
  If systemic or ocular diseases appear during the study, they will be followed up and observed for changes in retinal fiber layer thickness and macular thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Nakhoul Fa Nakhoul, MD, Principal Investigator — Baruch Padeh Medical Center
Locations (1):
- Baruch Padeh Medical Center, Poria – Neve Oved, Lower Galeli, Israel